CLINICAL TRIAL: NCT04805281
Title: Wear Behavior of Milled Posterior Crowns Fabricated From the New Gradient Technology Monolithic Zirconia 5Y-TZP/3Y-TZP Compared to Lithium Disilicate: (Randomized Clinical Trial)
Brief Title: Wear Behavior of Milled Posterior Crowns Fabricated From the New Monolithic Zirconia 5Y-TZP/3Y-TZP Compared to Lithium Disilicate
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Noran El-sharkawi, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 201020
Record Dates: First submitted 2021-02-17; First posted 2021-03-18 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Posterior Teeth; Worn Posterior Teeth; Endodontically Treated Teeth; Crowned Posterior Teeth
MeSH Terms: conditions — Tooth, Nonvital

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lithium Disilicate IPS e.max crowns in posterior teeth (Active Comparator)
  Interventions: Other: Lithium Dislicate IPS e.max crown
- Monolithic Zirconia (5Y-TZP/3-YTZP) crowns in posterior teeth (Experimental)
  Interventions: Other: monolithic zirconia (5Y-TZP/3-YTZ) ZirCAD Prime.

INTERVENTIONS:
Other: monolithic zirconia (5Y-TZP/3-YTZ) ZirCAD Prime. — wear of the new material of monolithic zirconia (5Y-TZP/3-YTZ) ZirCAD Prime in posterior teeth
  Arms: Monolithic Zirconia (5Y-TZP/3-YTZP) crowns in posterior teeth
Other: Lithium Dislicate IPS e.max crown — wear of lithium disilicate IPS e.max crown in posterior teeth
  Arms: Lithium Disilicate IPS e.max crowns in posterior teeth

SUMMARY:
In-vitro studies do not represent the actual masticatory environment and cannot simulate the intricate chewing pattern. Hence, there is a need for an in vivo study evaluating the wear potential of the newly introduced strength - color gradient multilayered zirconia IPS e.max ZirCAD Prime (5Y-TZP/3Y-TZP) and compare it to Lithium Disilicate IPS e.max CAD which has proven to have favorable wear patterns.

DETAILED DESCRIPTION:
* There will be no difference in wear caused by monolithic Zirconia (5Y-TZP/3Y-TZP) IPS E-max ZirCad Prime and Lithium Disilicate IPS e.max CAD to the antagonist.
* There will be no difference in the wear of the new monolithic zirconia IPS e.max ZirCAD Prime and lithium disilicate IPS e.max CAD.

ELIGIBILITY:
Inclusion Criteria:

* All subjects are required to:

  1- Be aged 21-50 years old, be able to read and sign the informed consent document. 2- Psychologically and physically able to withstand conventional dental procedures.

  3- Patients with mutilated posterior teeth indicated for full coverage restorations.

  4- Patients with sound natural antagonists. 5- Able to attend punctually for preplanned visits and evaluation. 6- Have no active periodontal or pulpal diseases.

  7- There should be no apparent loss or wear in opposing enamel.

Exclusion Criteria:

1. Patient with active resistant periodontal diseases.
2. Patients with parafunctional habits and bruxism.
3. Patients with poor oral hygiene, high caries risk and uncooperative patients. 3- Pregnant women.
4. Patients in the growth stage with partially erupted teeth. 5- Psychiatric problems or unrealistic expectations.

6- Lack of opposing dentition in the area of interest. 7- Restored occlusal surface opposing the planned restoration. 8- The presence of a removable or fixed orthodontic appliance.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
The amount of occlusal wear in natural antagonist enamel caused by the restorative material | 1 year
  The amount of occlusal wear in natural antagonist enamel, using digital superimposition of model scans after 1 year, measured in micrometer.

SECONDARY OUTCOMES:
The amount of occlusal wear in the restorative material itself | 1 year
  The amount of occlusal wear in the restorative material itself, using digital superimposition of model scans after 1 year, measured in micrometers.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No